CLINICAL TRIAL: NCT03514277
Title: Combined Administration of Bupivacaine and Exparel Versus Bupivacaine or Exparel Alone for Postoperative Analgesia in Posterior Lumbar Spine Surgery - A Prospective Randomized Study
Brief Title: A Prospective Study to Compare Bupivacaine and Exparel Versus Bupivacaine or Exparel Alone for Postoperative Pain Relief
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI decision to close study early
Sponsor: Virtua Health, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: VirtuaHealthExparel
Record Dates: First submitted 2018-03-15; First posted 2018-05-02 (Actual); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Low Back Pain; Lumbosacral Radiculopathy; Lumbar Disc Degeneration; Lumbar Disc Herniation; Stenosis; Spondylolisthesis; Spondylolysis; Deformity of Spine
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Constriction, Pathologic; Spondylolisthesis; Spondylolysis | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Local infiltration of EXPAREL and Bupivacaine (Active Comparator)
  Interventions: Drug: Exparel; Drug: Bupivacaine
- Local infiltration of Exparel (Active Comparator)
  Interventions: Drug: Exparel
- Local infiltration of Bupivacaine (Active Comparator)
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Exparel — 1 level patients - 20 mL Exparel; 2 level patients - 20 mL Exparel diluted to 40 mL
  Arms: Local infiltration of EXPAREL and Bupivacaine; Local infiltration of Exparel
Drug: Bupivacaine — 30 mL bupivacaine 0.5% w/v solution
  Arms: Local infiltration of Bupivacaine; Local infiltration of EXPAREL and Bupivacaine

SUMMARY:
The purpose of this study is to collect information about how patients feel when doctors manage their pain after lumbar spine surgery using a combination of EXPAREL® and bupivacaine injected into the lumbar spine at the end of surgery, compared to the patients that doctors use only EXPAREL® or bupivacaine to manage their pain. This information will help doctors determine which approach works best for patients who will receive surgery in their lumbar spine in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older;
2. Primary indication is low back pain, lumbosacral radiculopathy, lumbar disc degeneration, lumbar disc herniation, stenosis, spondylolisthesis, spondylolysis, or deformity requiring surgical intervention;
3. Scheduled to undergo primary, 1 or 2 level, posterior lumbar laminectomy with or without fusion, discectomy with fusion, or fusion at Virtua Memorial Hospital;
4. Willing to provide informed consent, participate in study, and comply with study protocol.

Exclusion Criteria:

1. Hypersensitivity or allergy to local anesthetics;
2. Pregnant or contemplating pregnancy prior to surgery;
3. Previous surgery in lumbar spine (i.e. other than microdiscectomy);
4. Prior treatment for alcohol, recreational drug, or opioid abuse;
5. Serious spinal conditions (e.g. spinal cord compression, cauda equina syndrome, spinal infection, spinal tumor, spinal fracture, inflammatory or systemic spinal arthritis);
6. Surgery involving more than 2 vertebral levels;
7. Worker's compensation or personal injury related to lumbar spine (treatment outcomes may be affected by patient's personal interests [21]; could also run into potential issues with reimbursement).
8. Lactating women
9. Patients with end stage liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greenleaf, MD, Principal Investigator — Princpal Investigator
Locations (1):
- Virtua Memorial Hospital, Mount Holly, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Publish research findings in relevant peer-reviewed journal

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Local Infiltration of EXPAREL and Bupivacaine | Local Infiltration of Exparel | Local Infiltration of Bupivacaine
Started | 11 | 4 | 4
Completed | 11 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Local Infiltration of EXPAREL and Bupivacaine | Local Infiltration of Exparel | Local Infiltration of Bupivacaine | Total
Number analyzed (Participants) | 11 | 4 | 4 | 19
Age, Continuous [Mean (Full Range); unit: years] | 67.8 [52 to 77] | 72.3 [66 to 80] | 67.3 [54 to 74] | 68.6 [52 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 2 | 10
  Male | 5 | 2 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 5
  White | 7 | 2 | 2 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Postoperative Pain Score
Description: Wong-Baker pain faces scale of 0-no pain, to 10-extreme pain
Time Frame: last day of hospitalization, average of 3 days in hospital
Population: Data is not collected for one patient in the Local infiltration of EXPAREL and Bupivacaine group
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Local Infiltration of EXPAREL and Bupivacaine | Local Infiltration of Exparel | Local Infiltration of Bupivacaine
Number analyzed (Participants) | 10 | 4 | 4
units on a scale | 5.2 [3.0 to 7.6] | 4.2 [3.1 to 5.6] | 5.6 [4.4 to 6.7]

2. Secondary Outcome: Total Consumption of Opioids During Hospital Stay
Description: All opioid analgesics will be converted into oral mg morphine equivalent to determine the total dose of opioids
Time Frame: last day of hospitalization, average of 3 days in hospital
Population: Data is not collected for one patient in the Local infiltration of EXPAREL and Bupivacaine group
Measure: Mean (Full Range); unit: milligram
Arm/Group | Local Infiltration of EXPAREL and Bupivacaine | Local Infiltration of Exparel | Local Infiltration of Bupivacaine
Number analyzed (Participants) | 10 | 4 | 4
milligram | 106.1 [0 to 300] | 87.3 [4 to 202.5] | 46.1 [13.5 to 81]

3. Secondary Outcome: Mean Time to Achieve Physical Therapy Discharge
Description: Mean time to achieve physical therapy discharge criteria
Time Frame: last day of hospitalization, average of 3 days in hospital
Population: This data was not collected
Arm/Group | Local Infiltration of EXPAREL and Bupivacaine | Local Infiltration of Exparel | Local Infiltration of Bupivacaine
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Opioid Related Adverse Events
Description: Number of Participants with Opioid Related Adverse Events
Time Frame: last day of hospitalization, average of 3 days in hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Local Infiltration of EXPAREL and Bupivacaine | Local Infiltration of Exparel | Local Infiltration of Bupivacaine
Number analyzed (Participants) | 11 | 4 | 4
Participants | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Duration of patient's hospital stay, an average of three days
Arm/Group | Local Infiltration of EXPAREL and Bupivacaine | Local Infiltration of Exparel | Local Infiltration of Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/11 | 0/4 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Local Infiltration of EXPAREL and Bupivacaine (N=11) | Local Infiltration of Exparel (N=4) | Local Infiltration of Bupivacaine (N=4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
lethargy (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Unsteadiness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Constitpation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT03514277/Prot_SAP_000.pdf